CLINICAL TRIAL: NCT05248100
Title: Strengthening the Continuity of HIV Care in Tanzania With Economic Support: Phase I
Brief Title: Rudi Kundini, Pamoja Kundini: Phase I
Acronym: RKPK: Phase I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: Health for a Prosperous Nation (Other); Rasello (Industry); Management and Development for Health (Unknown); Ministry of Health, Tanzania (Other Government); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sandra McCoy, Associate Professor in Residence, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R01MH125746 (NIH); R01MH125746 (NIH)
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: HIV (Human Immunodeficiency Virus)
Keywords: Conditional Cash Transfers; Tanzania; People Living With HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants will not be told during the consent process that as part of the study there are intervention and control clinics. Laboratory staff analyzing viral load samples will be blind to intervention/control attribution.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conditional Cash Transfer (Experimental): Eligible and consenting participants living in an intervention health facility catchment area will receive the same standard of care HIV tracing and clinical services as control participants, plus the opportunity to receive a one-time incentive of 22,500 Tanzanian Shillings (TSH) (~$10), with half (11,250 TSH) delivered upon enrollment in the study and half delivered after confirmation of the completion of a clinical visit if within 90 days of study enrollment.
  Interventions: Behavioral: Conditional Cash Transfer
- Control (No Intervention): Eligible and consenting participants living in a control health facility catchment area will receive the standard of care HIV tracing and clinical services.

INTERVENTIONS:
Behavioral: Conditional Cash Transfer — The intervention is a one-time cash transfer of 22,500 Tanzanian Shillings (~$10), with half (11,250 TSH) delivered upon enrollment in the study and half delivered after confirmation of the completion of a clinical visit if within 90 days of study enrollment.
  Arms: Conditional Cash Transfer

SUMMARY:
This protocol describes a 2-arm cluster, randomized controlled trial designed to test the effectiveness of a conditional cash transfer on viral suppression at 6 months among people living with HIV infection (PLHIV) in Tanzania who have disengaged from HIV care. Randomization will take place at the clinic level (HIV primary care clinics). The comparison group receives standard of care standard of care HIV tracing services according to Tanzania's National Guidelines for the Management of HIV and the Ministry of Health to locate potential participants, including home based care (HBC) tracing of PLHIV who have disengaged from primary care, the provision of counseling to return to HIV care, and the offer to schedule an HIV primary care appointment on the spot. Eligible adult PLHIV disengaged from HIV care and living in an intervention facility catchment area will receive the same standard of care HIV tracing and clinical services as control participants, plus the opportunity to receive a one-time cash transfer incentive, conditional upon confirmed completion of a clinical visit if within 90 days of study enrollment. The primary endpoint is viral suppression (<1000 copies/ml) at 6 months after study enrollment.

DETAILED DESCRIPTION:
The overall objective of this study is to evaluate the effectiveness of a home visit plus one-time financial incentive on the proportion of out of care PLHIV with viral load suppression (<1000 copies/ml) at 6 months after study enrollment. We will use a cluster, randomized controlled trial design with a sample size of 20 PLHIV in each of the 32 health facility catchment areas (N=640 PLHIV total) to examine the effect of a home visit plus one-time financial incentive on the primary outcome of viral suppression at 6 months. The study will take place across Geita and Kagera Regions (Lake Zone) in Tanzania.

This study will follow standard of care HIV tracing services according to Tanzania's National Guidelines for the Management of HIV and the Ministry of Health to locate potential participants, including home based care (HBC) tracing of PLHIV who have disengaged from primary care, the provision of counseling to return to HIV care, and the offer to schedule an HIV primary care appointment on the spot. Eligible and consenting participants living in an intervention health facility catchment area will receive the same standard of care HIV tracing and clinical services as control participants, plus the opportunity to receive a one-time incentive of 22,500 TSH (~$10 USD), with half (11,250 TSH) delivered upon enrollment in the study and half delivered after confirmation of the completion of a clinical visit if within 90 days of study enrollment.

Primary Endpoint:

1. Viral suppression (<1000 copies/ml) at 6 months after enrollment

Secondary Endpoints:

1. Viral suppression at 12 months after enrollment
2. Durable viral suppression at 12 months after enrollment
3. Appointment attendance
4. Time to re-linkage to care
5. Mortality at 12 months after enrollment
6. Re-linkage to care at 12 months after enrollment
7. Retention at 6 and 12 months, defined as the proportion of PLHIV on antiretroviral therapy (ART) at 6 months after enrollment and 12 months after enrollment, respectively

ELIGIBILITY:
Inclusion Criteria:

1. PLHIV living in the catchment area of a study health facility;
2. Age 18 years or older;
3. Phone ownership OR phone consistent phone access;
4. Classified as lost to follow up (LTFU) from HIV care (not attended a clinic appointment for ≥28 days since last scheduled appointment);
5. Has had a clinic appointment within the last 24 months, and
6. Provides written informed consent for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
6-month Viral Suppression | 6 months
  The proportion of people living with HIV (PLHIV) retained in HIV primary care and with suppressed HIV viral load 6 months following study enrollment. The primary outcome is expressed as a binary variable, defined as PLHIV who are on ART and with sufficient HIV viral suppression (<1000 copies/ml, WHO's threshold for virologic failure in LMICs) versus not on ART or viral failure (≥1000 copies/ml).

SECONDARY OUTCOMES:
12-month Viral Suppression | 12 months
  The proportion of people living with HIV (PLHIV) retained in HIV primary care and with suppressed HIV viral load 12 months following study enrollment. The primary outcome is expressed as a binary variable, defined as PLHIV who are on ART and with sufficient HIV viral suppression (<1000 copies/ml, the World Health Organization (WHO) threshold for virologic failure in low- and middle-income countries (LMIC)) versus not on ART or viral failure (≥1000 copies/ml).
Durable 12-month Viral Suppression | 12 months
  The proportion of people living with HIV (PLHIV) with durable HIV viral suppression at 12 months after study enrollment months (either: 1) ≥2 assessments of viral load, taken from up to 6 months prior to study enrollment and up to and including 12 months following study enrollment (the recommended timing of immunologic monitoring for stable PLHIV on ART with viral suppression), or 2) ≥3 assessments if baseline viral load is >1000 copies/ml (the recommended timing of immunologic monitoring mandates an additional follow-up assessment 3 months and again at 12 months)
6-month Appointment Attendance | 6 months
  The proportion of scheduled visits that were completed during the 0-6 month period
12-month Appointment Attendance | 12 months
  The proportion of scheduled visits that were completed during the 0-12 month period
12-month Mortality | 12 months
  The cumulative incidence of mortality at 12 months after study enrollment
Incidence of viral suppression | 12 months
  The cumulative incidence of mortality at 12 months after study enrollment
Incidence of re-linkage to HIV care | 12 months
  The cumulative incidence of re-linkage to to HIV care at 12 months after study enrollment
Time to re-linkage to HIV care | 12 months
  Time for patients to re-link back to HIV care
6 month retention in care | 6 months
  The proportion of people living with HIV (PLHIV) on ART at 6 months after study enrollment (PEPFAR considers those not retained on ART to include those who died, disengaged from care, stopped ART, or had no evidence of care for ≥28 days after a missed visit. Participants not found after exhaustive tracing efforts to rule out silent transfers will be classified as not retained on ART)
12 month retention in care | 12 months
  The proportion of people living with HIV (PLHIV) on ART at 12 months after study enrollment (PEPFAR considers those not retained on ART to include those who died, disengaged from care, stopped ART, or had no evidence of care for ≥28 days after a missed visit. Participants not found after exhaustive tracing efforts to rule out silent transfers will be classified as not retained on ART)

CONTACTS AND LOCATIONS:
Overall Officials: Jingshen Wang, PhD, Principal Investigator — University of California, Berkeley
Locations (2):
- Tanzania (2):
  - Geita Region, Geita
  - Kagera Region, Kagera

IPD SHARING:
Plan to Share IPD: Yes
Provided upon request
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Access Criteria: Provided upon request

REFERENCES:
- [Derived] Kadota JL, Packel LJ, Mlowe M, Ulenga N, Mwenda N, Njau PF, Dow WH, Wang J, Sabasaba A, McCoy SI. Rudi Kundini, Pamoja Kundini (RKPK): study protocol for a hybrid type 1 randomized effectiveness-implementation trial using data science and economic incentive strategies to strengthen the continuity of care among people living with HIV in Tanzania. Trials. 2024 Feb 10;25(1):114. doi: 10.1186/s13063-024-07960-x. PMID 38336793
- [Derived] Kadota JL, Packel LJ, Mlowe M, Ulenga N, Mwenda N, Njau PF, Dow WH, Wang J, Sabasaba A, McCoy SI. Rudi Kundini, Pamoja Kundini (RKPK): study protocol for a hybrid type 1 randomized effectiveness-implementation trial using data science and economic incentive strategies to strengthen the continuity of care among people living with HIV in Tanzania. Res Sq [Preprint]. 2023 Dec 20:rs.3.rs-3315136. doi: 10.21203/rs.3.rs-3315136/v1. PMID 38196655